CLINICAL TRIAL: NCT00409240
Title: Multi-Targeted Cardiac Risk Intervention in Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Providence VA Medical Center (U.S. Federal Agency)
Collaborators: Sandra A. Daugherty Foundation (Other)
Responsible Party: Principal Investigator, Wen-Chih Wu, Staff Cardiologist, Providence VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1127912
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-03

CONDITIONS: Diabetes; Hypertension; Dyslipidemia
Keywords: Group Intervention; Pharmacotherapy; Behavioral Modification; Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MEDIC Intervention (Experimental): Receives pharmacist-led behavioral and pharmacologic group intervention for cardiac risk reduction
  Interventions: Other: MEDIC
- Usual Care (No Intervention): Patient continued on usual care

INTERVENTIONS:
Other: MEDIC — Multidisciplinary Education and Diabetes Intervention for Cardiac risk reduction (MEDIC; a pharmacist-led behavioral and pharmacologic intervention in groups.
  Arms: MEDIC Intervention

SUMMARY:
Our study intends to test the efficacy of pharmacist-led group interventions on a weekly basis for 4-weeks, then on a monthly basis for 5 additional months to achieve concomitant reductions in hemoglobin A1c, lipids and blood pressure.

DETAILED DESCRIPTION:
Our project intends to study the 6-month efficacy of a pharmacist-led group intervention program that simultaneously target diabetes, hypertension and dyslipidemia. We hypothesize that pharmacist-led group interventions on a weekly basis for 4-weeks then on a monthly basis for 5 additional months may achieve concomitant reductions in hemoglobin A1c, lipids and blood pressure. We are proposing a pilot randomized controlled study to test the efficacy and feasibility of this approach.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus,
* >18 years old,
* with a documented HbA1c more than 7.0%,
* an LDL cholesterol >100 mg/dl AND a blood pressure >130/80 mm Hg documented at least once in the medical records within the last 6 months, and
* willing to comply with the study interventions will be eligible for the study.

Exclusion Criteria:

* pregnancy,
* unable to attend the group sessions,
* disease conditions such as psychiatric instability (acutely suicidal, psychotic) or organic brain injury that preclude them from performing diabetes self-care,
* enrolled in the Providence VAMC's Telehealth program

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chih Wu, MD, Principal Investigator — Providence VAMC, Brown Medical School
Locations (1):
- Providence VAMC, Providence, Rhode Island, United States

REFERENCES:
- [Result] Cohen LB, Taveira TH, Khatana SA, Dooley AG, Pirraglia PA, Wu WC. Pharmacist-led shared medical appointments for multiple cardiovascular risk reduction in patients with type 2 diabetes. Diabetes Educ. 2011 Nov-Dec;37(6):801-12. doi: 10.1177/0145721711423980. Epub 2011 Oct 21. PMID 22021025

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Veterans of the Providence VA Medical Center were eligible for the study. Dates of recruitment period were 2007-2009.
Period: Overall Study
Arm/Group | MEDIC Intervention | Usual Care
Started | 53 | 50
Completed | 50 | 49
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDIC Intervention | Usual Care | Total
Number analyzed (Participants) | 50 | 49 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (10.7) | 67.2 (9.4) | 68.5 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 50 | 47 | 97
Region of Enrollment [Number; unit: participants]
  United States | 50 | 49 | 99

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Achieving Hemoglobin A1C Goal, LDL Cholesterol Goal, and Systolic Blood Pressure Goal From the Enrollment Until the End of the Study
Description: Hemoglobin A1C target was < 7% LDL cholesterol goal of < 100mg/dl or <70mg/dl for patients at high risk-current cardiovascular disease Systolic blood pressure goal of <130mm Hg
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | MEDIC Intervention | Usual Care
Number analyzed (Participants) | 50 | 49
participants
  Percentage achieving A1C of <7% | 40.8 | 20.4
  Percentage achieving LDL at goal | 82.0 | 65.3
  Percentage achieving systolic Blood Pressure < 130 | 58.0 | 32.7
  Percentage Achieving combined goal A1c, SBP, LDL | 16.0 | 4.1

ADVERSE EVENTS:
Time Frame: The time frame for adverse event reporting was the entire duration of the study.
Arm/Group | MEDIC Intervention | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/49
Other Adverse Events (participants affected / at risk) | 2/50 | 3/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MEDIC Intervention (N=50) | Usual Care (N=49)
Infection (Infections and infestations) | 0 | 1 — Infections
Hypoglycemia (Endocrine disorders) | 2 | 0 — hypoglycemia
Lung cancer surgery (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — lung cancer surgery
(General disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Only 1 in 5 patients responded to the invitation to join the study and was willing to participate, participants were mostly male veterans, and pharmacists had prescribing privileges in the VA and in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No